CLINICAL TRIAL: NCT05397626
Title: Biofeedback and Hydrogen Water as Treatments for Chronic Fatigue Syndrome
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stony Brook University (Other)
Collaborators: Natural Wellness Now Health Products (Unknown)
Responsible Party: Principal Investigator, Fred Friedberg, Principal Investigator, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AWD00002822
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Chronic Fatigue Syndrome
Keywords: Heart Rhythm Biofeedback; Hydrogen Water
MeSH Terms: conditions — Fatigue Syndrome, Chronic | interventions — Water

STUDY DESIGN:
Intervention Model Description: This clinical study involves three active intervention groups: group 1 receiving heart rhythm biofeedback alone, group receiving hydrogen water alone, and group 3 receiving both heart rhythm biofeedback and hydrogen water.
Who Masked: Outcomes Assessor
Masking Description: Each participant fill out online outcome forms that involve no interaction with the principal investigator or study staff, thus avoiding any staff-specific influence on online outcome forms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Heart Rhythm Biofeedback (Active Comparator): Heart rhythm biofeedback is a non-invasive physiological treatment that is administered via an app downloaded to personal smart phones. It involves participants attaching a wireless sensor to the ear that monitors heart rate that is displayed on the phone screen app. The participant is actively involved in modifying the heart biofeedback to achieve optimal levels of heart rate variability, an established indicator of health and well-being and a potential factor in chronic fatigue syndrome. The treatment lasts 8 weeks.
  Interventions: Dietary Supplement: Hydrogen Water; Combination Product: Combined treatment: Heart rhythm biofeedback plus hydrogen water
- Hydrogen Water (Active Comparator): Hydrogen pills are mixed in a water glass that is ingested up to 3 times a day for 8 weeks. The hydrogen supplement is intended to reduce oxidative stress and inflammation both of which are implicated in the pathophysiology of chronic fatigue syndrome. This is an 8 week treatment.
  Interventions: Behavioral: Heart Rhythm Biofeedback; Combination Product: Combined treatment: Heart rhythm biofeedback plus hydrogen water
- Combined treatment: Heart rhythm biofeedback plus hydrogen water (Active Comparator): This condition combines heart rhythm biofeedback and hydrogen water, as described above, which is intended to assess any additive or synergistic effects of the two treatments. This is an 8 week treatment.
  Interventions: Behavioral: Heart Rhythm Biofeedback; Dietary Supplement: Hydrogen Water

INTERVENTIONS:
Behavioral: Heart Rhythm Biofeedback — Heart rhythm biofeedback is a non-invasive intervention intended to improve heart rate variability and physical resilience that is often limited in chronic fatigue syndrome
  Arms: Combined treatment: Heart rhythm biofeedback plus hydrogen water; Hydrogen Water
Dietary Supplement: Hydrogen Water — Hydrogen water, if ingested daily over several weeks, may have antioxidant and anti-inflammatory effects in chronic fatigue syndrome
  Arms: Combined treatment: Heart rhythm biofeedback plus hydrogen water; Heart Rhythm Biofeedback
Combination Product: Combined treatment: Heart rhythm biofeedback plus hydrogen water — This treatment is intended to explore the possible additive or synergistic effects of combining heart rhythm biofeedback and hydrogen water.
  Arms: Heart Rhythm Biofeedback; Hydrogen Water

SUMMARY:
The aim of this 10-week pilot study is to explore the potential benefit of two recently developed non-invasive interventions, heart rate variability biofeedback (HRV-BF) and OTC supplement hydrogen water, for the symptoms of chronic fatigue syndrome (CFS). Symptom measures and heart monitoring information will be generated by this study. Given the lack of effective treatments in this illness, these two non-invasive home-based treatments may help patients feel and function better.

DETAILED DESCRIPTION:
The aim of this 10-week pilot study is to explore the potential benefit of two recently developed non-invasive interventions, heart rate variability biofeedback (HRV-BF) and over the counter (OTC) supplement hydrogen water, for the symptoms of chronic fatigue syndrome (CFS). Symptom measures and heart monitoring information will be generated by this study. Given the lack of effective treatments in this illness, these two non-invasive home-based treatments may help patients feel and function better.

Participants will be randomized to one of the three study condition, HRV-BF alone, hydrogen water alone or combined HRV-BF and hydrogen water. All interventions are home-based with no in person visits. All communications with participants will be via virtual call, phone call, email and land mail.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of chronic fatigue, chronic fatigue syndrome, or something similar. ages 18-65. - BMI>30.

Exclusion Criteria:

* Other major medical condition or regular medication that produces fatigue. No home computer or internet access. No smart phone.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2022-05-23 (Actual); Primary Completion 2023-05-23 (Estimated); Study Completion 2023-05-23 (Estimated)

PRIMARY OUTCOMES:
Fatigue Severity Scale | 8 weeks
  self-report measure of fatigue impact on functioning.Minimum value=1; Maximum value=7; Range: 1.00-7.00. High scores indicate more sever fatigue and a worse outcome.

SECONDARY OUTCOMES:
Short Form-36 Physical Function Subscale | 8 weeks
  Self-report measure of physical functioning. The short-form 36 physical function subscale is composed of ten items encompassing a hierarchical range of difficulties. Each item is scores on the basis of the limitations perceived by surveyed individuals. Item scores (1, 2, or 3) are summed to obtain a total score, which can then be scaled relative to its range. Higher scores indicate higher physical function.
Depression, Anxiety and Stress Scale | 8 weeks
  Self-report measure if depression, anxiety and stress symptoms. This 21 item stress measure contains three 7-item subscales: anxiety, depression and stress. Domain scores are calculated by summing all items in a domain and multiplying by two.
Brief Resilience Scale | 8 weeks
  This 6 item self-report scale focuses on how quickly an individuals bounces back and physically and emotionally exhausting events. 5 answer choices range from strongly disagree to strongly agree. Higher scores indicate higher resilience.

CONTACTS AND LOCATIONS:
Overall Officials: FRED FRIEDBERG, Phd, Principal Investigator — Stony Brook University
Locations (1):
- Fred Friedberg, Stony Brook, New York, United States